CLINICAL TRIAL: NCT00677027
Title: Dose Escalation Safety Study of MM-10-001
Brief Title: Dose Escalation Safety Study of MM-10-001 in Healthy Subjects
Status: Unknown | Phase: Phase 1 | Type: Interventional
Last Known Status: Active, not recruiting
Sponsor: GlycaNova Norge AS (Industry)
Collaborators: Centre for clinical studies, Bergen, Norway (Unknown)
Responsible Party: Tor Albrektsen, GlycaNova Norge AS
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Supportive Care
Other Study IDs: 1.2006.3622 (REK); 07/02312 (SLV)
Record Dates: First submitted 2008-05-09; First posted 2008-05-13 (Estimated); Last update posted 2008-05-13 (Estimated); Status verified 2008-05

CONDITIONS: Healthy
Keywords: Beta-glucan; immune system; Healthy subjects
MeSH Terms: interventions — Lentinan

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- 1 (Experimental)
  Interventions: Other: lentinan
- 2 (Placebo Comparator)
  Interventions: Other: placebo

INTERVENTIONS:
Other: lentinan — Five dose levels of escalating concentrations of the test substance will be tested during the study periode. All patients will recieve each dose, which is to be taken daily for two weeks.
  Arms: 1
Other: placebo — Placebo
  Arms: 2

SUMMARY:
The purpose of this study is to evaluate the safety of increasing doses of MM-10-001 and to determine the dose of MM-10-001 that enhances the immune system in normal healthy subjects.

DETAILED DESCRIPTION:
The drug substance to be studied is a powder produced from shiitake mushroom, containing beta-glucans. The purpose of this study is to evaluate the safety of increasing doses of MM-10-001 and to determine the dose of MM-10-001 that enhances the immune system in normal healthy subjects.

ELIGIBILITY:
Inclusion Criteria:

Healthy subjects of both genders, age > 45 years old will be eligible for study.

Exclusion Criteria:

Subjects who:

1. Fail to give written informed consent
2. Have BMI over or equal to 30 kg/m2
3. Use corticosteroids (including inhaled steroids) or NSAIDs anti-inflammatory drugs
4. Have uncontrolled hypertension (sitting diastolic blood pressure>95 mmHg)
5. Have on-going allergy or history of anaphylactic reaction
6. Have on-going allergen specific immunotherapy
7. Are immuno-compromised (HIV infected, cancer and other disease affecting the basal immune response)
8. Have chronic inflammatory disease
9. Have diabetes (type 1 or type 2)
10. Have chronic severe renal disease (creatinine outside normal range)
11. Have chronic severe liver disease (ASAT and/or ALAT more than two times the upper limit of the normal range)
12. Have known cardiac failure
13. Have recently (less than 6 months) experienced myocardial infarction
14. Have gastrointestinal diseases (chronic gastritis, IBD, etc.)
15. Have acute or chronic pancreatitis or impaired pancreatic function, or history of pancreatitis
16. Have been vaccinated within the last three months
17. Eat diet supplement NG24 beta-glucan
18. Eat shiitake cheese
19. Have systemic fungal infection
20. Have any clinical condition that renders them unfit to participate including known/suspected drug or alcohol abuse
21. Do not fully understand the content of the informed consent
22. Pregnant and lactating women or women of childbearing potential not using adequate contraception.

Min Age: 45 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 50 (Estimated)
Dates: Start 2008-02; Primary Completion 2008-06 (Estimated); Study Completion 2008-06 (Estimated)

PRIMARY OUTCOMES:
Blood safety parameters | every second week

SECONDARY OUTCOMES:
Cell mediated immune response and cytokine production | every second week

CONTACTS AND LOCATIONS:
Overall Officials: Snorre Ofjord, MD, Principal Investigator — Centre for clinical studies, Bergen, Norway
Locations (1):
- Centre for clinical studies, Bergen, Paradis, Norway